CLINICAL TRIAL: NCT06347523
Title: The Application of a Preoperative Rehabilitation Program Based on Virtual Reality (VR) Technology in Patients Undergoing Anterior Cruciate Ligament (ACL) Reconstruction
Brief Title: VR-Based Preoperative Rehabilitation Program for Patients Undergoing Anterior Cruciate Ligament (ACL) Reconstruction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The sample size is insufficient
Sponsor: First Affiliated Hospital of Shantou University Medical College (Other)
Responsible Party: Principal Investigator, Zeshan Chen, Nurse Researcher, First Affiliated Hospital of Shantou University Medical College
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FirstShantou
Record Dates: First submitted 2024-03-22; First posted 2024-04-04 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Anterior Cruciate Ligament (ACL) Reconstruction; Preoperative Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The experimental group will receive an enhanced preoperative rehabilitation program incorporating Virtual Reality (VR) technology
  Interventions: Procedure: The VR-based preoperative rehabilitation program;
- control group (Active Comparator): The control group will receive standard nursing care.
  Interventions: Procedure: standard nursing care,

INTERVENTIONS:
Procedure: The VR-based preoperative rehabilitation program; — Patients are provided with VR headsets for personalized pre-rehabilitation educational videos prior to surgery. These videos cover psychological counseling, nutritional advice, and exercise instructions. Additionally, patients engage in VR interactive functional training. After surgery, patients continue with VR technology interactive functional training and watch postoperative educational videos. This intervention is initiated upon the patient's admission and continues until their discharge.
  Other Names: Virtual Reality Rehabilitation Program, VR Pre-op Rehab, VR Rehab Program
  Arms: experimental group
Procedure: standard nursing care, — Patients in the control group receive traditional preoperative rehabilitation methods, which may include the following interventions: Joint exercises and rehabilitation exercises guided by a physical therapist. Written or verbal rehabilitation educational materials.
  Arms: control group

SUMMARY:
Between April 2, 2024, and October 1, 2024, a study will be conducted at the Department of Orthopedics in the First Affiliated Hospital of Shantou University Medical College involving 120 patients who will undergo anterior cruciate ligament reconstruction surgery. They will be randomly divided into two groups: an experimental group and a control group.

DETAILED DESCRIPTION:
The control group will receive standard nursing care, while the experimental group will receive an enhanced preoperative rehabilitation program incorporating Virtual Reality (VR) technology. This program will include patient assessments, personalized exercise prescriptions, and VR-based educational videos covering psychological support, nutritional guidance, and exercise instructions.

Patients in the experimental group will use VR headsets for preoperative and postoperative interactive training sessions, as well as for viewing postoperative educational videos. The intervention will start upon admission and will continue until discharge.

Primary outcome measures will include knee joint range of motion and the Lysholm knee function score. Secondary measures will encompass anxiety, depression, pain scores, activities of daily living, time to ambulation, postoperative complications, and patient satisfaction.

Statistical analysis will be conducted to compare outcomes between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Individuals eligible for inclusion in the study are those who undergo their initial anterior cruciate ligament (ACL) reconstruction surgery, aged between 18 and 60 years, possess adequate hearing and vision, have clear consciousness, and demonstrate proficient language communication skills.

Exclusion Criteria:

* Individuals with cognitive impairments, severe hearing or vision impairments, limb paralysis, or non-compliance with the experiment will be excluded from participation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
knee joint range of motion | through study completion, an average of 6 months
  This refers to the bending of the knee joint, bringing the heel toward the buttocks
Lysholm knee function score | through study completion, an average of 6 months
  The Lysholm knee function score typically includes a series of questions or items that ask the patient to rate their ability to perform various activities and movements involving the knee joint. These activities may include walking, running, squatting, climbing stairs, and other functional tasks. Patients are asked to rate their knee function and any associated symptoms such as pain or instability.
  The scoring system for the Lysholm knee function score can vary, but it often ranges from 0 to 100, with higher scores indicating better knee function and lower scores suggesting greater impairment or limitations.

SECONDARY OUTCOMES:
SAS self-rating anxiety scale scale | through study completion, an average of 6 months
  The SAS scale typically consists of 20 items that assess both psychological and physical symptoms of anxiety, such as nervousness, restlessness, tension, and palpitations. Individuals are asked to rate how often they have experienced each symptom over a specific period, often the past week or two weeks. Responses are typically scored on a Likert scale, where higher scores indicate a greater degree of anxiety symptom severity.
  The total score on the SAS scale provides an overall measure of an individual's anxiety level. Higher scores indicate a higher level of anxiety, while lower scores suggest a lower level of anxiety.
SDS self-rating depression scale scale | through study completion, an average of 6 months
  The SDS scale typically consists of 20 items that assess various aspects of depression, including mood, sleep patterns, appetite changes, and physical symptoms. Individuals are asked to rate how often they have experienced each symptom over a specific period, often the past week or two weeks. Responses are typically scored on a Likert scale, where higher scores indicate a greater degree of depression symptom severity.
  The total score on the SDS scale provides an overall measure of an individual's depression level. Higher scores suggest a higher level of depressive symptoms, while lower scores indicate a lower level of depressive symptoms.
Visual Analog Scale pain score | through study completion, an average of 6 months
  The VAS pain score consists of a horizontal or vertical line, typically 10 centimeters in length. One end of the line is labeled "No Pain," indicating the absence of pain, while the other end is labeled "Worst Pain Imaginable," signifying the most severe pain imaginable.
  Assessment: Patients or study participants are asked to mark a point on the line that represents their current level of pain. The distance from the "No Pain" end to the marked point is measured in millimeters, and this measurement is recorded as the pain score.
  Scoring: The VAS pain score is recorded as a number on a scale from 0 to 10, where 0 indicates no pain, and 10 represents the worst possible pain. Higher scores correspond to higher perceived pain intensity.
Barthel Index for basic activities of daily living | through study completion, an average of 6 months
  The Barthel Index (BI) is a widely used tool for assessing an individual's level of independence in performing basic daily life activities. It comprises a series of tasks, such as eating, bathing, dressing, toileting, transferring from bed to chair, walking, and climbing stairs, among others. Each task is scored based on the individual's level of independence in completing it.
  Total Score: The total score on the Barthel Index is calculated by summing the scores for each task. Typically, the maximum score is 100, indicating complete independence in all assessed activities.
time to first ambulation post-surgery | through study completion, an average of 6 months
  it aims to assess when patients start moving after surgery, whether it's independent walking or with some degree of assistance.

OTHER OUTCOMES:
postoperative complications | through study completion, an average of 6 months
  Postoperative complications include any unexpected medical conditions or events that arise in a patient after surgery. These complications can include infections, bleeding, organ dysfunction, adverse reactions to anesthesia or medications, wound problems, and other health-related issues.
nursing satisfaction | through study completion, an average of 6 months
  Nursing satisfaction involves evaluating how content and fulfilled nursing staff or healthcare providers are with their professional roles, workplace conditions, and the support they receive. It measures their overall sense of well-being and job satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Yongsong Chen, Study Director — First Affiliated Hospital of Shantou University Medical College
Locations (1):
- "The First Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Scope of Data: The shared IPD will include participants' demographic information, ACL injury characteristics, treatment plans, recovery progress, and complication records.
  Data Format: The shared de-identified individual participant data will be provided in Excel format.
  Access Procedures: Access to the data will be granted through the submission of a data request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available within a specified period after the publication of primary results, within 6 to 12 months
Access Criteria: Research Purpose: only those planning further analysis or validation studies related to the original trial would qualify for data access.
  Data Request Procedure: Access seekers must submit their requests through a designated data request procedure. This procedure may require them to provide detailed information such as research plans, data utilization strategies, and anticipated outcomes.